CLINICAL TRIAL: NCT06756126
Title: A Multicenter, Open Label Phase II Clinical Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of AK120 in Adolescents With Moderate-to-severe AD
Brief Title: A Clinical Study of AK120 in Adolescents With Moderate-to-severe Atopic Dermatitis (AD)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK120-208
Record Dates: First submitted 2024-12-25; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK120 300mg every two weeks (Q2W) subcutaneous injection (Experimental): Subjects with heavy weight
  Interventions: Drug: AK120
- AK120 300mg every three weeks (Q3W) subcutaneous injection (Experimental): Subjects with light weight
  Interventions: Drug: AK120

INTERVENTIONS:
Drug: AK120 — AK120 subcutaneous injection

SUMMARY:
This is a A multicenter, open label, phase II clinical study to evaluate the safety, pharmacokinetics (PK), pharmacodynamics(PD), and preliminary efficacy of AK120 in adolescents with moderate-to-severe atopic dermatitis

DETAILED DESCRIPTION:
This is a A multicenter, open label, phase II clinical study aimed to evaluate the safety, PK, PD, and preliminary efficacy of AK120 in adolescents with moderate-to-severe AD. The entire study include screening period(week -4 to week 0), treatment and follow-up period(16 weeks). The duration of the study is about 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥12 <18 years old.
* Weight≥30kg at baseline.
* AD diagnosed at least half a year before screening.
* Subject with EASI score ≥16, IGA ≥ 3, BSA ≥ 10% at screening and baseline.

Exclusion Criteria:

* Acute onset of AD in 4 weeks prior to enrollment.
* Undergone or planned surgery during the study period within the 4 weeks prior to enrollment, or unable to fully recover from surgery before enrollment.
* Previously suffered from vernal keratoconjunctivitis (VKC) or atopic keratoconjunctivitis (AKC).
* Received systemic traditional Chinese medicine treatment within the 4 weeks before randomization or topical traditional Chinese medicine treatment within 1 week before randomization.
* Received treatment with other clinical study drugs within 1 month or 5 half-lives before randomization (whichever is longer).
* Have a history of allergies to any component of AK120 and/or severe allergic reactions to monoclonal antibodies.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events(AE) | week -4 to week 16
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.

SECONDARY OUTCOMES:
PK evaluation: maximum plasma concentration (Cmax) | Baseline till last follow-up visit ( up to day 113)
  Assessment of Cmax after AK120 administration.
PK evaluation: time to maximum plasma concentration (Tmax) | Baseline till last follow-up visit ( up to day 113)
  Assessment of Tmax after AK120 administration.
PD evaluation: Thymus and activation regulated chemokine (TARC)/CCL17 | Baseline till last follow-up visit ( up to day 113)
  Percentage change in TARC/CCL17 compared to baseline.
Change in Eczema Area and Severity Index (EASI) scores | week 0/2/4/8/12/16
  Percentage change in EASI scores from baseline.
Change in affected Body Surface Area (BSA) scores | week 0/2/4/8/12/16
  Percentage change in BSA score from baseline.
Subjects who achieved 0/1 in the Investigator's Global Assessment (IGA) | week 0/2/4/8/12/16
  Percentage of subjects who achieved IGA 0/1.
Change in Children's Dermatology Life Quality Index (CDLQI) scores | week 0/2/4/8/12/16
  Percentage change in CDLQI score from baseline.
Change in Patient Oriented Eczema Measure (POEM) scores | week 0/2/4/8/12/16
  Percentage change in POEM score from baseline.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Dongguan People's Hospital, Dongguan, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The University of Hong Kong - Shenzhen Hospital, Shenzhen, Guangdong
  - Hunan Pediatric Medical Union, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Ning Bo No.2 Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No